CLINICAL TRIAL: NCT00088517
Title: Whole Body Study of [11C]NNC-112 PET Imaging of Dopamine D1 Receptors
Brief Title: Positron Emission Tomography Imaging of Dopamine Receptors Using the Tracer [11C]NNC-112
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040170; 04-M-0170
Record Dates: First submitted 2004-07-27; First posted 2004-07-28 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-03

CONDITIONS: Healthy
Keywords: Biodistribution; MIRD; Radiation Absorbed Dose; Healthy; Prefrontal Cortex; Radiation Exposure; PET; Dopamine D1 Receptor; (11C)NNC-112; Healthy Volunteer; HV

INTERVENTIONS:
Drug: [11C]NNC-112

SUMMARY:
This study will investigate the use of [11C]NNC-112 in positron emission tomography (PET) scanning. PET is a technique that uses radioactive isotopes called tracers to provide images of the brain. Injected into the body, the isotopes lose their "radioactive strength" over time, sending out rays that can be picked up and "seen" by special detectors connected to a computer. The computer then makes a picture of the brain. This study will examine the distribution in the body of a new tracer called [11C]NNC-112.

Healthy normal volunteers between 18 and 70 years of age may be eligible for this study. Candidates are screened with a physical examination and blood and urine tests, including a urine drug screen. Women up to age 55 also have a pregnancy test.

Participants have a PET scan using the [11C]NNC-112 tracer. For this procedure, a catheter (small plastic tube) is placed into a vein in the subject's arm for injecting the tracer. Then, the subject lies on the scanner bed. After a preliminary "transmission scan," the tracer is injected, and PET scans are taken from the head to the upper thigh over a period of about 2 hours to show the distribution of radioactivity in the body. Blood pressure, breathing rate, and heart rate are checked before and after injection of the tracer, and blood and urine samples are collected after the PET scan.

DETAILED DESCRIPTION:
Abnormalities in dopaminergic neurotransmission have been implicated in several neurodegenerative and psychiatric disorders, such as Parkinson's disease, schizophrenia, attention-deficit-hyperactivity disorder and drug dependence. Among the Dopamine (DA) receptors, D1 receptors are understood to be involved in the regulation of motor and cognitive activity by modulating DAergic function. Neuroreceptor imaging with Positron Emission Tomography (PET) and Single Photon Emission Computerized Tomography (SPECT) allows in vivo quantification of the density and distribution of D1 receptors in humans. Recently, a new and superior PET radioligand for in vivo quantification of D1 receptors in extrastriatal regions has been developed. [11C]NNC-112 is a D1 radiotracer with high specific to nonspecific binding, making it suitable for imaging low density D1 receptors in extrastriatal regions such as the neocortex. Several studies in humans have confirmed the potential of this radiotracer, however, to date, dosimetry studies of [11C]NNC-112 in humans have not been performed.

The specific objective of this protocol is to estimate radiation-absorbed doses of [11C]NNC-112 in human subjects. For this purpose, we propose to perform a kinetic whole body imaging study of [11C]NNC-112 in healthy human subjects. We hypothesize that the level of radiation-absorbed doses of [11C]NNC-112 in humans will be within limits, and consequently, we should be able to move to the next stage of our imaging research, where we will use this radioligand to measure the density and distribution of D1 receptors in Parkinson's disease.

ELIGIBILITY:
INCLUSION CRITERIA

All subjects must be healthy and aged 18-70 years.

EXCLUSION CRITERIA

Current psychiatric disease, substance abuse or severe systemic disease based on history and physical exam

Laboratory tests with clinically significant abnormalities

More than moderate hypertension

Any prior participation in other research protocols within the past year that involve radiation, with the exception of plain radiography studies (i.e., chest x-rays).

Pregnancy and Breast Feeding

Positive HIV test

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 2004-07; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Abi-Dargham A, Martinez D, Mawlawi O, Simpson N, Hwang DR, Slifstein M, Anjilvel S, Pidcock J, Guo NN, Lombardo I, Mann JJ, Van Heertum R, Foged C, Halldin C, Laruelle M. Measurement of striatal and extrastriatal dopamine D1 receptor binding potential with [11C]NNC 112 in humans: validation and reproducibility. J Cereb Blood Flow Metab. 2000 Feb;20(2):225-43. doi: 10.1097/00004647-200002000-00003. PMID 10698059
- [Background] Abi-Dargham A, Mawlawi O, Lombardo I, Gil R, Martinez D, Huang Y, Hwang DR, Keilp J, Kochan L, Van Heertum R, Gorman JM, Laruelle M. Prefrontal dopamine D1 receptors and working memory in schizophrenia. J Neurosci. 2002 May 1;22(9):3708-19. doi: 10.1523/JNEUROSCI.22-09-03708.2002. PMID 11978847
- [Background] Andersen PH, Gronvald FC, Hohlweg R, Hansen LB, Guddal E, Braestrup C, Nielsen EB. NNC-112, NNC-687 and NNC-756, new selective and highly potent dopamine D1 receptor antagonists. Eur J Pharmacol. 1992 Aug 14;219(1):45-52. doi: 10.1016/0014-2999(92)90578-r. PMID 1397049